CLINICAL TRIAL: NCT01567943
Title: Novel EtG-Based Contingency Management for Alcohol in the Severely Mentally Ill
Brief Title: Contingency Management of Alcohol Abuse in the Severely Mentally ILL
Acronym: CMETG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Richard Ries, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41552-G
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Alcohol Abuse; Schizophrenia; Bipolar Disorder; Major Depressive Disorder
Keywords: alcohol abuse; drug abuse; schizophrenia; bipolar disorder; major depressive disorder; contingency management; psychosocial treatment
MeSH Terms: conditions — Alcoholism; Schizophrenia; Bipolar Disorder; Depressive Disorder, Major; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contingency Management (Experimental): Contingency Management plus treatment as usual
  Interventions: Behavioral: Contingency Management
- Non-contingent control group (No Intervention): Treatment as usual plus reinforcement for attendance

INTERVENTIONS:
Behavioral: Contingency Management — Behavioral reinforcement for alcohol abstinence
  Arms: Contingency Management

SUMMARY:
The investigators will evaluate the efficacy of a comprehensive 12-week contingency management intervention for treating alcohol dependence for persons with severe mental illness who are seen within the context of a community mental health center setting. The primary contingency will be submission of alcohol-free urines. Additional reinforcers will be provided for intensive outpatient addiction treatment attendance. Reinforcers will be vouchers or actual items useful for day-to-day living. Participants will be 120 adults diagnosed with alcohol dependance and severe mental illness.

DETAILED DESCRIPTION:
The contingency management (CM) paradigm that will be used is the variable magnitude of reinforcement procedure. In order to encourage engagement in study procedures and reduce dropout in the randomized sample, all participants will undergo a 4-week pre-randomization induction period. During the induction period, participants will be reinforced for providing urine-tests three times a week. Those who demonstrate study participation and need for treatment during the induction period will be randomized to receive treatment as usual and either 1) 12 weeks of CM for alcohol abstinence (assessed by Ethyl glucuronide immunoassay urine-test) AND weekly reinforcement for intensive outpatient addiction treatment attendance; or 2) 12 weeks of reinforcement for providing urine-samples and continued study involvement. Randomization will be used to assign participants to treatment conditions.

The primary outcome will be changes in alcohol use assessed by Ehyl glucuronide immunoassay urine-tests, breath-tests, as well as self- and clinician-reported alcohol use. The secondary outcome will be changes in intensive outpatient group attendance assessed by intensive outpatient clinician-report, as well as administrative data sources, and self-report. Other outcomes will include: urine-tests and self-reported illicit drug use, psychiatric symptoms, other outpatient treatment utilization, HIV-risk, and nicotine use. All outcomes will be assessed [for 4-weeks prior to study enrollment (self-report, clinician ratings etc)] and throughout the 4-week induction, 12-week intervention, and 3-month follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Currently receiving psychiatric [AND intensive outpatient addiction treatment] at Community Psychiatric Clinic (CPC).
2. Aged 18 to 65 years.
3. Ability to understand written and spoken English language.
4. DSM-IV diagnosis of alcohol dependence as assessed by the MINI psychiatric interview.
5. Diagnosis of current serious mental illness: schizophrenia, schizoaffective disorders, bipolar disorder I or II, or recurring major depressive disorders as assessed by the MINI psychiatric interview.
6. Alcohol use in the month prior to study entry: self-reported alcohol use of 5 days or more during the 30 days prior to study entry (5 drinking days/month is selected based on previous research reporting alcohol use in 18% of days assessed in a sample of psychiatric outpatients with co-occurring SUDs & SMI).120
7. A CPC treating clinician must affirm the potential participant is safe to participate in the study.

Exclusion Criteria:

1. A significant risk of dangerous alcohol withdrawal: a history of alcohol detoxification or seizure in the last 12 months AND participant or clinician concern that abstinence will induce dangerous alcohol withdrawal.
2. DSM-IV diagnosis of current (last year) drug dependence as assessed by the MINI interview.
3. Any medical/psychiatric condition, or severity of that condition, that in the opinion of the PI, would compromise safe study participation.
4. Chart defined organic brain disorder or dementia.
5. Inability to provide informed consent as measured by the University of California San Diego Brief Assessment of Capacity to Consent (UBACC), a tool designed to screen for ability to provide informed consent for research. If indicated by the UBACC screening process, the more comprehensive MacCAT-CR will be used.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-03; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Ries, MD, Principal Investigator — University of Washington; Michael McDonell, PhD, Principal Investigator — Washington State University
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 123 participants were enrolled, but only 79 met criteria to be randomized. Criteria for randomization included: EtG-positive urine sample during 4-week pre-randomization phase of the study, and adequate attendance during the pre-randomization phase.
Groups:
- Pre-randomization Drop-out: These participants were enrolled/consented in the study but not randomized to the Contingency Management or Control conditions.
Period: Overall Study
Arm/Group | Contingency Management | Non-contingent Control Group | Pre-randomization Drop-out
Started | 40 | 39 | 44
Completed | 26 | 29 | 44
Not Completed | 14 | 10 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contingency Management | Non-contingent Control Group | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 79
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.55 (9.92) | 46.23 (10.55) | 45.38 (10.24)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 26 | 24 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use as Assessed by Ethyl Glucuronide Detection in Urine
Description: Mean EtG value (in ng/mL). 150ng/mL or above = EtG-positive, 149ng/mL or below = EtG-negative. EtG = ethyl glucuronide, alcohol biomarker detectable in urine.
Time Frame: Over 16 weeks of treatment (repeated measure)
Measure: Mean (Standard Error); unit: EtG Value (nanograms per milileter)
Arm/Group | Contingency Management | Non-contingent Control Group
Number analyzed (Participants) | 40 | 39
EtG Value (nanograms per milileter) | 408.86 (39.57) | 734.79 (40.66)

2. Secondary Outcome: Change in Intensive Outpatient Substance Abuse Treatment Attendance
Time Frame: During 16 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of addiction tx attended
Arm/Group | Contingency Management | Non-contingent Control Group
Number analyzed (Participants) | 40 | 39
percentage of addiction tx attended | 57 (34) | 53 (37)

3. Secondary Outcome: Self Report Drug Use
Time Frame: through 7 months of study
Reporting Status: Not Posted

4. Secondary Outcome: Other Drug Use as Measured by Urinalysis
Time Frame: through 7 months of study
Reporting Status: Not Posted

5. Secondary Outcome: Community Outcomes
Description: (jail bookings, ER visits, mental health and substance abuse service utilization)
Time Frame: entire study period, and three month prior and after study involvement
Reporting Status: Not Posted

6. Secondary Outcome: Psychiatric Symptomology
Description: Brief Symptom Inventory; Positive and Negative Symptom Scale
Time Frame: throughout 7 months of study
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Contingency Management | Non-contingent Control Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No